CLINICAL TRIAL: NCT03429244
Title: PSMA-PET for Biopsy and Treatment Guidance in Primary Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Clinton Bahler, Assistant Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IUSCC-0658; 1802085219 (Other: Indiana University IRB)
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Results first posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 68Ga-PSMA-11 PET will be performed and we will study how the knowledge of the results helps inform treatment decisions.
Masking Description: Two separate Radiologists (one from Nuclear Medicine and one from MRI) will do the imaging reads in a blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prostate cancer- men being treated with radical prostatectomy (Experimental): Men being treated for prostate cancer with radical prostatectromy were enrolled in this arm.
  Interventions: Diagnostic Test: 68Ga-PSMA-11 PET-MRI
- Prostate cancer- men undergoing cancer screening or active surveillance (Experimental): Men undergoing cancer screening or active surveillance were enrolled in this arm.
  Interventions: Diagnostic Test: 68Ga-PSMA-11 PET-MRI
- Prostate cancer- focal therapy (Experimental): Men undergoing focal therapy with high intensity focused ultrasound are in this group.
  Interventions: Diagnostic Test: 68Ga-PSMA-11 PET-MRI

INTERVENTIONS:
Diagnostic Test: 68Ga-PSMA-11 PET-MRI — Patients will undergo injection of 68Ga-PSMA-11 at the time of pre-treatment MRI scan and followed until biopsy and/or surgical resection.

SUMMARY:
The overall objective of this Early Phase Clinical Trial is to begin defining the accuracy of 68Ga-PSMA-11 for detecting the location and size of clinically significant prostate cancer lesions in low and intermediate risk disease.

A molecularly-targeted probe (68Ga-PSMA-11), coupled with an advanced clinical imaging system (Siemens Biograph VisionPET-CT), will improve accuracy during biopsy and staging. We propose detailed intra-lesion whole-mount pathologic analysis as the gold standard for critically assessing PSMA PET accuracy in patients undergoing surgery, and blinded PSMA PET-CT comparison with standard multi-parametric MRI (mpMRI) for patients having biopsy on active surveillance. This intensive testing of the accuracy and value of PSMA-based tracers requires our unique collaboration of surgeons, radiologists, pathologists, and imaging scientists with decades of experience and innovation.

DETAILED DESCRIPTION:
This is a prospective, single arm, phase 2 clinical trial. This patient population will have low (1 = Gleason 3 + 3) or intermediate risk (2 = 3 + 4; 3 = 4 + 3) prostate cancer. It will also enroll those who are at high risk of significant prostate cancer (4Kscore >20%, SelectMDx >20%, PSA density >0.15). Patients will be scheduled for magnetic resonance imaging (MRI) as part of routine care for either surgical planning or for further biopsy. Following the informed consent process, patients who enroll in the study will receive a PSMA positron emission tomography (PET) study along with their standard of care (SOC) MRI on an integrated PET-MRI. Registration of PET and MRI will be done using software to generate the PET-MRI images. Patients receiving SOC MRI guided biopsy will receive additional PET guided biopsies as indicated in a single session. The sensitivity and specificity will be evaluated along with the ability of the tracer to inform the treatment planning. Patients receiving surgical removal of the prostate will have a slice-by-slice whole mount analysis to assess the sensitivity and specificity the PSMA PET.

Primary Objectives Define the accuracy of 68Ga-PSMA-11 PET-CT for detecting the clinically significant prostate cancer lesion.

Secondary Objectives Evaluate how knowledge of the PSMA-PET might inform treatment planning.

Exploratory Objectives Generate pilot data for future larger clinical trials

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Must provide written informed consent
3. Presence of low or intermediate risk prostate cancer or at risk of having intermediate risk cancer

   a. Intermediate risk prostate cancer: i. Grade group 2 = 3 + 4, or ii. Grade group 3 = 4 + 3 b. At Risk of intermediate risk prostate cancer: i. 4K score ≥ 20%, or ii. Select MDx ≥ 20%, or iii. PSA Density ≥ 0.15 iv. Grade group 1= 3+3 (iv. Note: Where multiple cancer lesions are present on biopsy, it is allowable to have Gleason 8 or 9 cancer lesions if they are in addition to the intermediate risk cancer as described above.)
4. Scheduled for MRI or has recently completed SOC MRI (within 6 months) for further biopsy, or surgical removal, or focal therapy.
5. Willing and able to lie still for approximately 50 minutes in an enclosed space for the CT.

Exclusion Criteria:

1. Participation in another investigational trial involving research exposure to ionizing radiation concurrently or within 30 days.
2. Does not meet safety criteria for MRI scan (e.g. metal implant that is not allowed).
3. Significant acute or chronic medical, neurologic, or psychiatric illness in the subject that, in the judgment of the Principal Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a prostate cancer study which can only be done with males.
Enrollment: 36 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Bahler, MD, Principal Investigator — Indiana University School of Medicine
Locations (4):
- United States (4):
  - Indiana University Health North Hospital, Carmel, Indiana
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Undecided
For multi-institutional projects with data sharing agreement.

REFERENCES:
- [Result] Bahler CD, Green MA, Tann MA, Swensson JK, Collins K, Alexoff D, Kung H, Brocken E, Mathias CJ, Cheng L, Hutchins GD, Koch MO. Assessing extra-prostatic extension for surgical guidance in prostate cancer: Comparing two PSMA-PET tracers with the standard-of-care. Urol Oncol. 2023 Jan;41(1):48.e1-48.e9. doi: 10.1016/j.urolonc.2022.10.003. Epub 2022 Nov 1. PMID 36333187

RESULTS

PARTICIPANT FLOW:
Groups:
- Prostate Cancer Being Treated With Radical Prostatectomy: 68Ga-PSMA-11 PET: Patients will undergo injection of 68Ga-PSMA-11 and PET scanning followed by surgical resection. The PET scan will be used to predict cancer grade, location, and stage and compared to final pathology as reference standard.
- Screening for Prostate Cancer or on Active Surveillance: This group gets PSMA-PET scan to help guide biopsy decision for initial diagnosis or active surveillance decisions.
- Prostate Cancer Being Treated With Focal Therapy: This group gets PSMA-PET scan to help inform focal therapy treatment decisions (HIFU hemiablation).
Period: Overall Study
Arm/Group | Prostate Cancer Being Treated With Radical Prostatectomy | Screening for Prostate Cancer or on Active Surveillance | Prostate Cancer Being Treated With Focal Therapy
Started | 16 | 11 | 9
Completed | 14 | 10 | 8
Not Completed | 2 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prostate Cancer Being Treated With Radical Prostatectomy | Screening for Prostate Cancer or on Active Surveillance | Prostate Cancer Being Treated With Focal Therapy | Total
Number analyzed (Participants) | 14 | 10 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (6.6) | 63.1 (6.5) | 66.5 (8.9) | 62.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 14 | 10 | 8 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 5
  White | 11 | 9 | 7 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 10 | 8 | 32
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (4.6) | 29.8 (5.4) | 29.8 (6.2) | 28.7 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy of PSMA PET
Description: Sensitivity and specificity for EPE using whole-mount analysis or biopsy pathology. EPE is extra-prostatic extension which means the cancer extends beyond the boundary of the prostate into adjacent muscle or fatty tissue.
Time Frame: 60 days
Population: 13 patients in this arm had imaging followed by surgery. Each patient contributed 2 sides. This primary outcome is only available for this treatment arm as the reference standard is only available for this treatment arm. That is, the other 2 treatment arms did not undergo prostatectomy with pathological evaluation.
Measure: Number; unit: percentage
Units Other Than Participants: Left and right nerve bundle
Groups:
- Prostate Cancer Being Treated With Radical Prostatectomy: 68Ga-PSMA-11 PET-MRI: Patients will undergo injection of 68Ga-PSMA-11 and PET scan followed by surgical resection.
Arm/Group | Prostate Cancer Being Treated With Radical Prostatectomy
Number analyzed (Participants) | 13
Number analyzed (Left and right nerve bundle) | 26
percentage
  Sensitivity for EPE (%) | 100
  Specificity for EPE (%) | 74

2. Secondary Outcome: Impact of PSMA PET-CT on Treatment Plan for Surgery or Biopsy
Description: Does the PSMA-PET change the treatment or biopsy decision. The surgeon will look at imaging prior to a procedure (prostatectomy, HIFU, or biopsy) to see if it informs the procedure steps. Does the imaging add new information about the cancer that could alter the biopsy or treatment? PSMA-PET scans were obtained in 3 different contexts as listed below (prior to prostate removal, screening for cancer or on active surveillance, and prior to focal therapy). We calculate the percentage of cases that had the treatment or followup plan altered by the investigational imaging agent.
  For example, if the PET imaging showed cancer was organ confined, then the surgeon may elect to increase the nerve sparing. For the active surveillance group, if this PET imaging showed a new lesion in the prostate, when compared to ultrasound or MRI, then the biopsy may have been altered to target this new lesion. For focal therapy, the treatment could be expanded to ensure any new PET lesions are covered.
Time Frame: 60 days
Population: Does the PET imaging help or inform or possibly help or inform the patient management?
Measure: Count of Participants; unit: Participants
Arm/Group | Prostate Cancer Being Treated With Radical Prostatectomy | Screening for Prostate Cancer or on Active Surveillance | Prostate Cancer Being Treated With Focal Therapy
Number analyzed (Participants) | 13 | 10 | 8
Participants | 10 | 8 | 5

ADVERSE EVENTS:
Time Frame: The patients were observed for adverse event at the time of investigational agent injection and PET scanning (within 60minutes of the scan).
Description: This variable is tracking adverse events at the scan event only as noted above.
Arm/Group | Prostate Cancer Being Treated With Radical Prostatectomy | Screening for Prostate Cancer or on Active Surveillance | Prostate Cancer Being Treated With Focal Therapy
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/14 | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT03429244/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT03429244/ICF_001.pdf